CLINICAL TRIAL: NCT06436014
Title: Evaluation of the Effect of Virtual Reality Application on Postoperative Pain and Anxiety in Women Aged 50-70 According to the Type of Surgery: A Randomized Controlled Trial
Brief Title: Evaluation of the Effect of Virtual Reality Application on Postoperative Pain and Anxiety in Women Aged 50-70
Acronym: Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Songul Gungor, Lecturer Phd, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OsmaniyeKorkutAtaUniversity
Record Dates: First submitted 2024-03-02; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pain Management After Surgery
Keywords: Virtual Reality (VR); Postoperative Pain; Pain Management Patient Experience
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group 1 ( Pre-Test + Intervention + Post-Test) (Participants undergoing total knee replacement surgery, subjected to pre-test followed by VR intervention) Group 2 (receiving only pre-test) Group 3 (Intervention Only + Post-Test) (Participants undergoing hysterectomy surgery, subjected to pre-test followed by VR intervention) Group 4 (Post-Test Only) (Participants undergoing hysterectomy surgery, receiving only pre-test)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Total Knee Replacement VR Intervention Group (Experimental): Pre-Test + Intervention + Post-Test) (Participants who underwent total knee replacement Participants who underwent total knee replacement surgery and received a pre-test, followed by VR intervention.Participants in this group are initially assessed with VAS and Beck Anxiety Scale.
  Subsequently, VR intervention is administered to this group. After the intervention, participants are reassessed with VAS and Beck Anxiety Scale.
  Interventions: Other: Providing VR experience
- Total Knee Replacement Control Group (No Intervention): Pre-Test (Participants who underwent total knee replacement surgery and received only a pre-test).Participants in this group are initially assessed with VAS and Beck Anxiety Scale.
- Hysterectomy VR Intervention Group (Experimental): Pre-Test + Intervention + Post-Test) Participants who underwent hysterectomy surgery and received a pre-test, followed by VR intervention.Participants in this group are initially assessed with a pre-test, followed by VR intervention.
  Interventions: Other: Providing VR experience
- Hysterectomy Control Group (No Intervention): Participants who underwent hysterectomy surgery and received only a pre-test).Participants are assessed only with VAS and Beck Anxiety Scale after the intervention period.

INTERVENTIONS:
Other: Providing VR experience — Participants undergoing VR intervention will experience a VR program of their choice based on personal preferences. Among these programs are videos offering natural visual experiences. For instance, participants can opt for videos featuring seaside views, forest tours, or lake landscapes.
  Arms: Hysterectomy VR Intervention Group; Total Knee Replacement VR Intervention Group

SUMMARY:
Surgical interventions, while significant milestones in patients' physical recovery processes, can be a major source of concern for patients due to postoperative pain, which is also an important component of postoperative care. If postoperative pain is not managed properly, it can lead to increased levels of anxiety and fear, as well as deterioration in overall comfort and quality of life. The ineffective management of postoperative pain has economic and medical consequences such as patient dissatisfaction, delayed hospital discharge, increased rates of hospital readmission, and dissatisfaction with medical care. Therefore, effective management of postoperative pain is of great importance for patient well-being. Factors associated with postoperative pain have been reported in many studies. For example, being female and the type of surgery. Therefore, considering gender and type of surgery in the management of postoperative pain is crucial to optimize the recovery process for patients. In recent years, research on the use of innovative technologies such as virtual reality in the management of postoperative pain has increased. Virtual reality can reduce postoperative pain by creating a sense of being in a different environment for patients and diverting their attention away from pain.

DETAILED DESCRIPTION:
Understanding the use of virtual reality applications in the medical field and their effects on pain perception and sensitivity in women is important. This study aims to evaluate the potential impact of virtual reality technology on pain and anxiety during the postoperative period in women aged 50-70. The research will be conducted at Osmaniye State Hospital. The general hypotheses of this study are that virtual reality application is effective in reducing postoperative pain and anxiety. The sub-hypotheses aim to determine the effect of virtual reality application among women undergoing two different types of surgeries (total knee replacement and hysterectomy). The method used in the research includes a randomized controlled trial design, involving application and control conditions across four different groups. Data will be collected through a questionnaire. The questionnaire will gather participants' demographic information, and their pain levels will be assessed using the Visual Analogue Scale (VAS) while their anxiety levels will be evaluated using the Beck Anxiety Scale. After the pre-test, virtual reality application will be administered to experimental groups with two different types of surgeries. No intervention will be applied to the control group before the post-test. Ethical approval and written informed consent will be obtained from the participants. Participants' postoperative pain and anxiety levels, analgesic usage amounts and frequencies will be recorded, and feedback related to their virtual reality experiences will be obtained. In the study, the rotation method will be used to randomly assign participants to experimental and control groups. The rotation method aims to place each patient sequentially into the next group. For example, the first patient undergoing total knee replacement surgery will be assigned to Group 1, and then the second patient undergoing total knee replacement surgery will be assigned to Group 2, the first patient undergoing hysterectomy surgery will be assigned to Group 3, and the second patient undergoing hysterectomy surgery will be assigned to Group 4. Thus, separate control and application groups will be formed for each type of surgery. This study is original and important as it will be the first study in our country to evaluate the impact of virtual reality on pain and anxiety in 50-70-year-old women according to the type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 50-70,
* Being female,
* Having adequate vision and hearing,
* Having American Society of Anesthesiologists (ASA) physical status classification I and II,
* Undergoing elective total knee replacement or hysterectomy surgery,
* Having a similar analgesia protocol,
* Being on the first postoperative day,
* Scoring 5 or higher on the Visual Analogue Scale (VAS) assessment,
* Being able to speak and understand Turkish.

Exclusion Criteria:

* Having chronic pain,
* Scoring below 5 on the Visual Analogue Scale (VAS) assessment,
* Experiencing vertigo or motion-sensitive nausea,
* Being diagnosed with severe anxiety by a specialist physician,
* Having claustrophobia,
* Having head or neck conditions that prevent wearing virtual reality goggles,
* Having a Glasgow Coma Score <15,
* Having psychiatric, cognitive, or neurological impairments,
* Having visual or hearing impairments.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women aged 50-70 years
Enrollment: 76 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The VR application is effective in changing postoperative pain. | The researcher's first visit to the patient on postoperative day 1.
  Pretest with VAS is administered on the first postopera tive day to women aged 50-70 undergoing total knee replacement and hysterectomy. • Subsequently, VR intervention is conducted. • Following the intervention, participants are re-evaluated with VAS.

SECONDARY OUTCOMES:
The VR application is effective in changing postoperative anxiety. | The researcher's first visit to the patient on postoperative day 1.
  Pretest with Beck Anxiety Scale is administered on the first postoperative day
  to women aged 50-70 undergoing total knee replacement and hysterectomy. • Subsequently, VR intervention is conducted. • Following the intervention, participants are re-evaluated with Beck Anxiety Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Songül GÜNGÖR, Phd, Principal Investigator — Osmaniye Korkut Ata University; Ayşe TAŞTEKİN, associate professor, Study Director — Afyonkarahisar Health Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Osmaniye Korkut Ata University, Merkez, Osmani̇ye
  - Osmaniye State Hospital, Merkez, Osmani̇ye